CLINICAL TRIAL: NCT02218632
Title: Galactosaemia, a Modifiable Multi-system Glycosylation Disorder?
Brief Title: Glycosylation in Patients With Galactosaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's University Hospital, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other); Medical Research Charities Group Ireland (Unknown); University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12020; grant PAC number 12.64 (Other Grant/Funding Number: MRCG/HRB)
Record Dates: First submitted 2014-08-07; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Classical Galactosaemia
Keywords: Galactosaemia; Dysglycosylation; Diet
MeSH Terms: conditions — Galactosemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lactose-free diet (Active Comparator): lactose-free diet (standard therapy) vs. lactose-free diet plus temporary oral galactose supplements
  Interventions: Other: lactose-free diet
- lactose free diet (Active Comparator): lactose-free diet (standard therapy)
  Interventions: Dietary Supplement: Temporary oral galactose supplements

INTERVENTIONS:
Other: lactose-free diet — standard diet
  Other Names: On established lactose-free diet
  Arms: lactose-free diet
Dietary Supplement: Temporary oral galactose supplements — galactose supplements in the range of physiological galactose production
  Other Names: In addition to lactose-free diet
  Arms: lactose free diet

SUMMARY:
Galactosaemia is an inherited condition caused by a lack of an enzyme (catalyst) which normally breaks down galactose (the sugar found in milk products). This affects 1:19,000 births annually in Ireland (the highest incidence worldwide) and is screened for by the National Newborn Screening Programme. When an affected infant is diagnosed, galactose is immediately restricted from the diet. This prevents often fatal liver disease and other immediate complications. However, despite early treatment the majority of affected patients go on to develop long-term complications such as intellectual impairment, neurological complications, speech difficulties and infertility in females. The underlying mechanisms for these complications are unclear. The investigators have shown in detailed biochemical and gene analysis studies that major abnormalities affecting the function of complex molecules in the body, particularly glycoproteins, (consisting of sugar chains attached to proteins) persist in treated individuals which may lead to disturbances of the body's intrinsic cellular machinery and relate to the complications seen.

In this research the investigators expand on from their earlier studies to see if they can identify biomarkers and parts of the galactose/glycosylation pathways which could be modified or changed with new treatments to improve outcomes for this condition (i.e., IgG N glycans).

In more detail, the investigators test the use of the most abundant glycoprotein in human plasma (IgG) as an improved clinical test for monitoring the galactose control needed in patients and also to see if some patients (including children aged 5-12 yrs) might have a better predicted outcome with moderate increases of galactose in the diet. The investigators believe that these studies greatly improve the understanding of Galactosaemia with a view to improving current treatment options and future outcomes.

DETAILED DESCRIPTION:
Classical Galactosaemia is an inherited disorder of galactose metabolism caused by profound deficiency of galactose-1-phosphate uridyltransferase (GALT: EC 2.7.712). This results in a systemic accumulation of toxic galactose intermediates and a decrease in the level of UDP-galactose, a required sugar for glycosylation. Galactosaemia has a relatively high incidence in Ireland, (1:19,000 births) presenting a particular public health problem. The neonatal life-threatening phenotype (liver disease, coagulopathy and sepsis) is rescued by restriction of dietary galactose. However, outcomes of treatment are disappointing beyond the neonatal period (even after successful newborn screening, early treatment and long term compliance). The majority of Irish patients harbour the severe Q188R Galt mutation.

56.5% of Irish patients ≥ 6yrs have IQs ≤ 79; and 91.2% of Irish female patients ≥ 13yrs have Premature Ovarian Insufficiency (POI). Unfortunately, the basic pathophysiology of this condition remains enigmatic with limited treatment approaches.

In their earlier work, the investigators reported very considerable variation in patient outcomes, even among siblings. The investigators have proposed that these differences are determined by variation in galactose accessory pathways (beyond the GALT deficiency). This may result in variable galactose tolerance in patients with linked variation in glycosylation pathways which could allow for enhanced UDP-galactose bioavailability essential for glycosylation. In their previous and current work the investigators have identified ongoing dysregulation of glycoprotein formation and expression of genes involved in glycan biosynthesis and cell signalling pathways in treated Galactosaemia patients.

The present proposal, which builds on published previous work, enables the investigators to establish that Galactosaemia is a modifiable, multi-systemic glycosylation defect. The overall objectives of the work are to progress the development of biochemical markers (IgG N-glycan analysis) as prognostic indices for potentially modifiable relevant pathways. The investigators consider how the phenotype could be relaxed in some patients with Classical Galactosaemia, initially by studies of modification of exogenous galactose requirements to identify if the ongoing glycan processing defects identified may be improved reflecting accessory pathways of galactose disposal.

Study Aim: Expand previous and published work using IgG N-glycan analysis to examine the glycosylation status of treated adult Galactosaemia patients in a larger study and develop this test as a reliable diagnostic tool. The investigators also carry out a pilot study to examine the effects of diet relaxation in paediatric patients (5-12 yrs) aiming to determine optimum galactose intake levels for this cohort with the hope of preventing long-term complications later in life. The investigators propose that this research offers new insights into the ongoing pathophysiology of this rare disorder with the possibility of developing new treatment targets, which over time could be cost-effective by preventing major disability.

ELIGIBILITY:
Inclusion Criteria:

* Classical galactosaemia
* Q188R Genotype
* On lactose-free diet
* No complications, condition well controlled
* Male/femal adults and children aged between 5-12 yrs.
* Informed consent /assent
* Patient attend the Galactosaemia Clinic, NCIMD Dublin

Exclusion Criteria:

* Complications, such as cataracts
* Galactosaemia varaint, no Q188R-Genotype
* Poor compliance
* Intercurrent illness
* Individual may not complete follow up
* Children below 5 years of age
* Unable to provide informed consent
* Patient not under the care of Galactosaemia Clinic, NCIMD Dublin

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with Classical Galactosaemia on a lactose-free diet in Ireland with disease specific complications | 2 years
  clinical monitoring and biochemical assessment to determine the number of patients with classical galactsaemia in Ireland with disease specific complications

SECONDARY OUTCOMES:
Number of participants with Classical Galactosaemia with variations in their glycosylation status in the Irish cohort | 2 years
  Glycosylation analysis: IgG N-glycan analysis (serum test)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Treacy, MD, Prof, Principal Investigator — University Children's Hospital Dublin Irleland
Locations (1):
- National Centre for Inherited Metabolic Disorders, Children's University Hospital, Temple Street, Dublin, Ireland

REFERENCES:
- [Result] Coss KP, Hawkes CP, Adamczyk B, Stockmann H, Crushell E, Saldova R, Knerr I, Rubio-Gozalbo ME, Monavari AA, Rudd PM, Treacy EP. N-glycan abnormalities in children with galactosemia. J Proteome Res. 2014 Feb 7;13(2):385-94. doi: 10.1021/pr4008305. Epub 2013 Dec 20. PMID 24359113
- [Result] Knerr I, Coss KP, Doran PP, Hughes J, Wareham N, Burling K, Treacy EP. Leptin levels in children and adults with classic galactosaemia. JIMD Rep. 2013;9:125-131. doi: 10.1007/8904_2012_191. Epub 2012 Nov 7. PMID 23430559